CLINICAL TRIAL: NCT01173718
Title: Evaluation of the GORE® ACUSEAL Vascular Graft for Hemodialysis Access (ACUSEAL, AVG 08-06)
Brief Title: Evaluation of the GORE® ACUSEAL Vascular Graft for Hemodialysis Access
Acronym: ACUSEAL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVG 08-06
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Results first posted 2013-07-02 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: End Stage Renal Disease
Keywords: Hemodialysis; Vascular Graft
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GORE® ACUSEAL Vascular Graft (Experimental)
  Interventions: Device: GORE® ACUSEAL Vascular Graft

INTERVENTIONS:
Device: GORE® ACUSEAL Vascular Graft — Surgical implantation of the GORE® ACUSEAL Vascular Graft for Hemodialysis per the Investigator's standard of practice.

SUMMARY:
This study is a prospective, non-randomized, multi-center evaluation of the performance of the GORE® ACUSEAL Vascular Graft. The study will enroll patients with End-Stage Renal Disease (ESRD), who are either currently receiving or expected to require hemodialysis through a prosthetic vascular graft within 30 days. Gore proposes to demonstrate that the 6 month cumulative patency of the GORE® ACUSEAL Vascular Graft is similar to that of other arteriovenous grafts (AVGs). > >>

>

>> A total of 138 Subjects will be enrolled. Once the study procedure has been successfully completed, cannulation may occur at any time at the Investigator's discretion. >

>>

>

>> Subjects will be selected from up to 20 Investigational Sites.

ELIGIBILITY:
Inclusion Criteria:>

1. Patient requires the creation of a vascular access graft for hemodialysis secondary to a diagnosis of End-Stage Renal Disease. >

   >>
2. Patient is currently on hemodialysis or ready to begin hemodialysis within 30 days following placement of study device. > >>
3. The patient must be able to have the vascular access graft placed in an upper extremity. >

   >>
4. The patient is 18 years of age or older. >

   >>
5. The patient has a reasonable expectation of remaining on hemodialysis for 12 months. >

   >>
6. The patient or his/her legal guardian understands the study and is willing and able to comply with follow-up requirements. > >>
7. The patient or his/her legal guardian is willing to provide informed consent. >

   >>

   >

   >>

   >

   >> Exclusion Criteria:>

   >>

<!-- -->

1. The patient has a documented and unsuccessfully treated ipsilateral central venous stenosis via imaging technique.>

   >>
2. The patient currently has a known or suspected systemic infection.>

   >>
3. The patient has a known hypercoagulable or bleeding disorder or requires treatment with warfarin or heparin.>

   >>
4. The patient has had a previous instance of Heparin Induced Thrombocytopenia type 2 (HIT-2) or has known sensitivity to heparin. >

   >>
5. The patient is being considered for a live (living donor either related or unrelated to patient) donor kidney transplant.>

   >>
6. The patient is enrolled in another investigational study.>

   >>
7. The patient has co-morbid conditions that may limit their ability to comply with study and follow-up requirements.>

   >>
8. Study device is intended to be used temporarily.>

   >>
9. The patient has had >2 previous arteriovenous accesses in treatment arm.>

   >>
10. Patient is taking Aggrenox®.>

    >>
11. The patient is in need of, or is scheduled for a different vascular surgical procedure within 30 days of the study procedure.>

    >>
12. The patient is currently taking maintenance immunosuppressant medication such as rapamycin, mycophenolate or mycophenolic acid, prednisone(>10 mg), cyclosporine, tacrolimus or cyclophosphamide.>

    >>
13. The patient has a known hypercoagulable or bleeding disorder or requires treatment with warfarin or heparin.>

    >>
14. Life expectancy is less than 12 months.>

    >>
15. The patient is pregnant.>

    >>
16. The patient is a poor compliance risk (i.e. history of IV or oral drug abuse).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2010-07; Primary Completion 2012-09 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Glickman, MD, Principal Investigator — Sentara Vascular Specialists

REFERENCES:
- [Derived] Glickman MH, Burgess J, Cull D, Roy-Chaudhury P, Schanzer H. Prospective multicenter study with a 1-year analysis of a new vascular graft used for early cannulation in patients undergoing hemodialysis. J Vasc Surg. 2015 Aug;62(2):434-41. doi: 10.1016/j.jvs.2015.03.020. Epub 2015 May 4. PMID 25953016

RESULTS

PARTICIPANT FLOW:
Groups:
- GORE® ACUSEAL Vascular Graft: GORE® ACUSEAL Vascular Graft : Surgical implantation of the GORE® ACUSEAL Graft for Hemodialysis per the Investigator's standard of practice.
Period: Overall Study
Arm/Group | GORE® ACUSEAL Vascular Graft
Started | 138
Completed | 94
Not Completed | 44
Not completed — Death | 17
Not completed — Abandonment of study graft | 27

BASELINE CHARACTERISTICS:
Arm/Group | GORE® ACUSEAL Vascular Graft
Number analyzed (Participants) | 138
Age Continuous [Mean (Standard Deviation); unit: years] | 63 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 67
Region of Enrollment [Number; unit: participants]
  United States | 138

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Patency at 6 Months
Description: Percentage of subjects free from loss of access for hemodialysis at the study access site, assessed at 6 month.
Time Frame: 6 Months
Population: All subjects with unknown cumulative patency status at the 6 month window were omitted from calculations
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GORE® ACUSEAL Vascular Graft
Number analyzed (Participants) | 128
percentage of participants | 83.6 [76 to 89.5]

2. Primary Outcome: Freedom From Bleeding at 6 Months
Description: Percentage of subjects free from both major and minor bleeding events, assessed at 6-months
Time Frame: 6 Months
Population: All subjects with unknown bleeding status at the 6 month window were omitted from calculations
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GORE® ACUSEAL Vascular Graft
Number analyzed (Participants) | 113
percentage of participants | 87.6 [80.1 to 93.1]

3. Secondary Outcome: Primary Unassisted Patency at 6 Months
Description: The primary unassisted patency is defined as the percentage of subjects free from the first occurence of either access thrombosis or an access procedure performed to maintain access patency.
Time Frame: 6 Months
Population: All subjects with unknown primary unassisted patency status at the 6 month window were omitted from calculations
Measure: Number; unit: percentage of participants
Arm/Group | GORE® ACUSEAL Vascular Graft
Number analyzed (Participants) | 131
percentage of participants | 45 [37.6 to 54.6]

4. Secondary Outcome: Time to Event Analysis (Cumulative Patency)
Description: The cumulative patency at 6 months and time-to-loss of cumulative patency will be estimated using the Kaplan-Meier survival curve for time-to-event analysis to obtain estimates accounting for censoring.
Time Frame: 6 Months
Population: All subjects with unknown time to event analysis (cumulative patency) status at the 6 month window were omitted from calculations
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GORE® ACUSEAL Vascular Graft
Number analyzed (Participants) | 128
percentage of participants | 84.2 [76.8 to 89.4]

5. Secondary Outcome: Time to First Cannulation
Description: The time to first cannulation is defined as the time from access placement to the first cannulation of the GORE® ACUSEAL Vascular Graft.
Time Frame: Time of access placement to first cannulation, assessed up to one week
Population: All subjects with unknown time to first cannulation at the 6 month window were omitted from calculations
Measure: Number; unit: percentage of grafts
Arm/Group | GORE® ACUSEAL Vascular Graft
Number analyzed (Participants) | 135
percentage of grafts
  Cannulated within 24 hours of procedure | 22.2
  Cannulated within 48 hours of procedure | 35.6
  Cannulated within 72 hours of procedure | 40.0
  Cannulated within 1 week of procedure | 51.9

6. Secondary Outcome: Time to Potential Central Venous Catheter Removal
Description: The time to potential central venous catheter removal is defined as the time from the initial study procedure to the third consecutive cannulation through the GORE® ACUSEAL Vascular Graft in which hemodialysis is carried out. The third consecutive cannulation is a surrogate endpoint for time to CVC removal. Typically, CVC removal is ordered after the third consecutive cannulation.
Time Frame: Initial study procedure to the third consecutive cannulation, assessed from day 3 thru day 123
Population: All subjects with unknown time to potential central venous catheter removal at the 6 month window were omitted from calculations
Measure: Median (Full Range); unit: days
Arm/Group | GORE® ACUSEAL Vascular Graft
Number analyzed (Participants) | 134
days | 15.5 [3 to 123]

ADVERSE EVENTS:
Groups:
- GORE® ACUSEAL Vascular Graft: GORE® ACUSEAL Vascular Graft
Arm/Group | GORE® ACUSEAL Vascular Graft
Serious Adverse Events (participants affected / at risk) | 74/138
Other Adverse Events (participants affected / at risk) | 0/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GORE® ACUSEAL Vascular Graft (N=138)
Anemia (Blood and lymphatic system disorders) | 6 (6)
Anemia aggravated (Blood and lymphatic system disorders) | 1 (1)
Chronic thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (3)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 3 (3)
Cardiac arrhythmia (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Congestive heart failure (Cardiac disorders) | 4 (4)
Coronary artery disease (Cardiac disorders) | 1 (1)
Diastolic heart failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Non ST segment elevation myocardial infarction (Cardiac disorders) | 1 (1)
Non STEMI (Cardiac disorders) | 4 (4)
Non-sustained ventricular tachycardia (Cardiac disorders) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1)
STEMI (Cardiac disorders) | 1 (1)
SVT (Cardiac disorders) | 1 (1)
Unstable angina (Cardiac disorders) | 2 (2)
Polycystic kidney (Congenital, familial and genetic disorders) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1)
Erosive esophagitis (Gastrointestinal disorders) | 1 (1)
GI bleed (Gastrointestinal disorders) | 3 (3)
Gastric polyps (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal bleed (Gastrointestinal disorders) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 2 (4)
Ileitis (Gastrointestinal disorders) | 1 (1)
Large intestine mass (Gastrointestinal disorders) | 1 (1)
Peptic ulcer disease (Gastrointestinal disorders) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Edema extremity upper (General disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Multi organ failure (General disorders) | 1 (1)
Swelling arm (General disorders) | 1 (1)
Liver failure (Hepatobiliary disorders) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1)
Arteriovenous graft site cellulitis (Infections and infestations) | 1 (1)
Arteriovenous graft site infection (Infections and infestations) | 9 (10)
Bacterial endocarditis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Cellulitis of hand (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Community acquired pneumonia (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 1 (1)
Graft infection (Infections and infestations) | 1 (1)
Hematoma infection (Infections and infestations) | 1 (1)
Incision site infection (Infections and infestations) | 1 (1)
Infected toe (Infections and infestations) | 1 (1)
Peripheral gangrene (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7)
Pyelonephritis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 4 (4)
Septic shock (Infections and infestations) | 2 (2)
Septicemia (Infections and infestations) | 2 (2)
Staphylococcal bacteremia (Infections and infestations) | 1 (1)
Staphylococcus aureus bacteremia (Infections and infestations) | 2 (2)
Staphylococcus epidermidis infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3)
Urinary tract infection pseudomonal (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Wound infection due to staphylococcus aureus (Infections and infestations) | 1 (1)
Anastomotic ulcer hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Arteriovenous graft site hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Bleeding of suture site (Injury, poisoning and procedural complications) | 1 (1)
Burst fracture (Injury, poisoning and procedural complications) | 1 (1)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Pulseless (Investigations) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Volume overload (Metabolism and nutrition disorders) | 2 (2)
Hand pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colonic neoplasm NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastrointestinal stromal tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Multiple myeloma progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anoxic encephalopathy (Nervous system disorders) | 1 (1)
CVA (Nervous system disorders) | 3 (4)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Encephalopathy acute (Nervous system disorders) | 1 (1)
Ischemic neuropathy (Nervous system disorders) | 2 (2)
Stroke (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Acute confusional state (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 4 (6)
End stage renal disease (ESRD) (Renal and urinary disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercapnic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Renal transplant (Surgical and medical procedures) | 2 (2)
Critical limb ischemia (Vascular disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Hypertension worsened (Vascular disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (2)
Hypertensive urgency (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 5 (7)
Peripheral ischemia (Vascular disorders) | 1 (1)
Peripheral vascular disease (Vascular disorders) | 1 (1)
Steal syndrome (Vascular disorders) | 15 (15)
Uncontrolled hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Gore has the right to review disclosures, requesting a delay of less than 90 days. Each investigator will postpone single center publications until after disclosure of multi-center data, less than 12 months from study completion/termination at all participating sites.